CLINICAL TRIAL: NCT00128999
Title: A Phase I/II Dose Escalation Study Using Induction Chemotherapy and Intensity-Modulated Radiation Therapy Guided by Combined CT and PET Imaging for Patients With Non-Small Cell Lung Cancer
Brief Title: Study Using Induction Chemotherapy and Intensity-Modulated Radiation Therapy Guided by Combined CT and PET Imaging for Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alberta Health services (Other)
Organization: AHS Cancer Control Alberta (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LU-11-0035
Record Dates: First submitted 2005-08-09; First posted 2005-08-11 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2007-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: radiation therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Intensity-Modulated Radiation Therapy

SUMMARY:
Lung cancer is the leading cause of cancer-related mortality in the United States (US) and Canada. Because of the high incidence and mortality of this disease, small improvements in the management of this disease translates into large numbers of patients having improved outcomes after treatment. Radiation therapy is widely used to treat patients with lung cancer. However, the radiation dose to the tumor has been limited by the proximity of normal structures to the tumor, such as the lung, the spinal cord and the esophagus. The normal structures must not be exposed to excessive radiation doses. A new technique, called intensity-modulated radiotherapy delivers radiation to tumors such that the normal structures around the tumor are exposed to less radiation than previously achievable. This technique is already used to treat head and neck cancers. This study will use this technique to deliver more intensified radiation to the lung tumor after the patient receives two cycles of chemotherapy. A new imaging technique, called positron emission tomography (PET), has been found to be more sensitive and specific at detecting the extent of the tumor in the lung than the older imaging technique of computed tomography (CT). This study will use both the PET and CT to target the radiation beams. Following treatment, the patients will be followed up to assess the side effects of normal tissues and response of the tumor to the treatment.

DETAILED DESCRIPTION:
Hypothesis and Objectives: The hypothesis that respiratory gated IMRT can escalate safely radiation doses for NSCLC with induction chemotherapy will be tested. The intent of the study is to determine the maximum tolerable dose of radiotherapy for NSCLC, using a novel treatment planning technique with accelerated fractionation, given with state-of-the-art imaging guidance.

Primary Objective:

* To establish the maximum tolerated dose of radiotherapy by assessing treatment toxicity according to the acute RTOG grading scale.

Secondary Objectives:

* To evaluate the treatment toxicity of the combination regimen according to the chronic RTOG grading scale;
* Quality of Life: to be assessed using the EORTC QLQ-C30 and LC13;
* To determine progression-free survival with this regimen;
* To identify partial organ tolerance doses for lung, esophagus and heart.

Schema and Methods: Eligible patients who have consented will receive two cycles of cisplatin-vinorelbine chemotherapy. Thoracic radiotherapy will be given afterwards according to the dose-escalating scale. Only one dose level will open at one time. Dose level 1: 84. Gy in 35 fractions over 7 wks; Dose level 2: 79.5 Gy in 40 fractions over 6 wks; Dose level 3: 75. Gy in 40 fractions over 5 wks.

Eligibility Criteria:

* Patients with histologically-proven, by biopsy or cytology, unresected NSCLC
* Patients with AJC Stage I-III if all detectable tumors can be encompassed by radiation therapy fields
* Patients with positive supraclavicular node (N3) or malignant pleural effusion are not eligible.
* Age >= 18
* Karnofsky performance status >= 70
* ANC > 1.5; Plt > 100,000; Hct > 30%; AST (SGOT) < 1.5 ULN; serum creatinine < 1.5 mg/dL
* Patients must have measurable disease on the CT and PET images
* Patients must have a FEV1 > 1.0 L
* Evaluation of the total lung volume receiving 20 Gy (V20) must be < 30%; mean esophageal dose must be < 32 Gy; and the esophageal V 55 < 28%.
* Patients must have a satisfactory IMRT plan prior to start of radiotherapy.

Statistical Considerations

Primary Endpoint: The frequency of patients developing unacceptable (grade 3 or higher) toxicity according to the RTOG acute toxicity scale attributable to radiotherapy. Acute radiotherapy toxicities are defined as those toxicities that occur within 90 days from the start of radiotherapy.

Sample Size: In order to establish the maximum tolerated dose (MTD) of radiotherapy that can be delivered using IMRT following induction chemotherapy, acceptable morbidity criteria must be defined. Based on the Radiation Therapy Oncology Group (RTOG) 94-10, the dose limiting toxicity (DLT: defined as a grade 3 or 4 non-hematologic toxicity) rate for this study is determined to be 40%. After 7 evaluable patients have been followed for a minimum of 90 days from the start of radiation therapy, patients will be evaluated with respect to treatment morbidity. If there are no acute dose limiting toxicities in the first 5 patients (0/5), then the current dose will be deemed to be acceptable and will be escalated. If there is 1 acute DLT observed in the first 5 patients (1/5) and no acute DLTs in the last two patients (0/2), then the dose will be deemed to be acceptable and will be escalated. Otherwise the current dose will be deemed to be too toxic and escalation will end. This design gives at least 90% confidence that the true acute DLT rate at a given dose level is less than 40% and for any given dose level, the probability of not escalating when the true toxicity rate is 40% or higher is at least 88%.

Safety Monitoring and Stoppage Rules: An SAE is any untoward medical occurrence that:

* results in death;
* is life-threatening (patient is at immediate risk of death);
* requires inpatient hospitalization or prolongation of existing hospitalization;
* results in persistent or significant disability/incapacity;
* is congenital anomaly/birth defect;
* important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the patient and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

Reporting of SAEs is as follows:

1. Complete the Serious Adverse Event Report;
2. Fax the Serious Adverse Event Report within 24 hours of the investigator's or designee's knowledge of the event to the attention of: Dr. Wilson Roa (780) 432-8517 (tel);(780) 432-8380 (fax) and Dr. Don Yee (403) 944-2895 (tel);(403) 283-1651 (fax);
3. Accrual may be stopped immediately as indicated upon review and confirmation of the SAE by the two PIs.

Recruitment and Reporting: The projection rate of accrual was based on a previous preliminary study. At this rate, it would take three months to complete accrual for each of the 3 dose levels. A three-month waiting period is required prior to dose escalation to the next level. Hence, an estimate of 7 months is conservatively allowed for each level, amounting to a total of 21 months to complete accrual, treatments and waiting period for the primary endpoint. The first manuscript on this study will be completed by the end of two years. Analysis for the reporting treatment results will contain tabulation of all cases entered and any excluded from analysis, with reasons for the exclusion. Respective institutional accrual and observed endpoints of MTD, toxicity, progression-free survival and quality of life will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III
* Unresectable non-small cell lung cancer (NSCLC)
* EEV1 equal to or greater than 1.0L

Exclusion Criteria:

* Positive supraclavicular noce (N2) or malignant pleural effusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5
Dates: Start 2003-09; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
safety and adverse effects

SECONDARY OUTCOMES:
efficacy and survival

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Roa, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada